CLINICAL TRIAL: NCT00539877
Title: Phase I Study of Interperitoneal Chenotherapy in Patients With Gastric Adenocarainoma With Peritoneal Seeding
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-05-017
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Stomach Neoplasms
Keywords: Gstric cancer; Pritoneal seeding; Intraperitoneal chemotherapy; Irinotecan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irinotecan — Postoperative day 1, IP CPT-11 chemotherapy will be given by CAPD catheter. CPT-11 in 1L of normal saline, prewarmed to 37°C will be given intraperitoneally.
  If there is no DLT and patients agree with the treatment, patients can receive 3 more times of IP chemotherapy with same dose of CPT-11 at 3 weeks interval. After total 4 cycles of IP chemotherapy, peritoneal disease will be reassessed with abdominal-pelvis CT. Pharmacokinetic study is not planned with this treatment.

SUMMARY:
Stomach cancer is the most common cancer, and is still leading cause of death in Korea. Peritoneal seeding is the most common metastases of gastric cancer, and is the most frequent cause of death from this disease. In addition, there is no standard treatment for peritoneal dissemination. Even though systemic intravenous chemotherapy is the standard treatment for metastatic stomach cancer at present, it does not improve the survival of patients with peritoneal dissemination. Because intraperitoneal(IP) administration results in high concentration locally with low systemic toxicity, clinical investigators have confirmed the safety and pharmacokinetic advantage associated with IP delivery of a number of antineoplastic agents with known activity in cancer. In ovarian cancer, a large randomized trial demonstrated a small but statistically and clinically significant survival advantage for women receiving a portion of their therapy intraperitoneally. Drugs such as 5-fluorouracil, cisplatin, mitomycin-C, paclitaxel and docetaxel are used for IP chemotherapy in patients with gastric cancer. Even the small number of phase III trials reported, some studies showed improvement in survival for patients randomized to IP therapy compared to those receiving no postoperative treatment. Irinotecan(7-ethyl-10-[4-(1-pipperidino)-1-piperidino] carbonyloxy camptothecin; CPT-11), clinically effective in the treatment of colorectal, lung and gastric cancer, is a carbamate prodrug metabolized to its active metabolite, 7-ethyl-10-hydroxycamptothecin (SN-38). In mouse model, IP administration of CPT-11 was significantly more effective than intravenous administration for control of both peritoneal seeding and liver metastasis. However, phamacokinetics of CPT-11 with peritoneal administration in human beings is not well studied. Although Japanese investigators reported pharmacokinetic data of CPT-11 with few patients, there is no data about maximum tolerated dose of CPT-11 intraperitoneally.

DETAILED DESCRIPTION:
Objectives : The objectives of this study are to assess the feasibility, to determine the maximum tolerated dose, and to assess the toxicities of intraperitoneally administered CPT-11 in gastric cancer patients with peritoneal seeding.

Methods : This is open-labeled, non-randomized phase I study in the patients eligible for the following criteria. Patients more than 18 years old with gastric adenocarcinoma, histologically proven, will be enrolled at the time of surgery, and the signed informed consent will be obtained prior to surgery. Preoperative studies should have resectable advanced disease. The operative finding and biopsy of suspected peritoneum must show peritoneal involvement of adenocarcinoma. The subjects should not have any previous chemotherapy, immunotherapy or radiotherapy and any major biological abnormalities. Prior to the initiation of study, patient will receive palliative gastrectomy(total or subtotal) and has a CAPD catheter. Postoperative day 1, IP chemotherapy will be given by CAPD catheter. For dose level 1, CPT-11(provided by CJ Pharmaceutical Company) 50mg/m2 in 1L of normal saline, prewarmed to 37°C will be given intraperitoneally. Plasma samples will be collected prior IP chemotherapy, and samples of plasma, peritoneal fluid and urine will be obtained at 0.5, 1.5, 2, 3.5, 8, 12, and 25.5, 49, 56 hours following chemotherapy. Three patients will be accrued to each dose level. If none of these three patients experienced a dose-limiting toxicity (DLT), the dose will be increased in a subsequent group of three patients to 100 mg/m2.If one of the first three patients experienced DLT, three more patients will be accrued to that dose level. If none of these additional three patients experienced DLT, then the dose will be escalated. If one of the additional three patients experienced DLT, then either an additional cohort of patients could be added or escalation terminated. If two or more of the second group of three patients experienced DLT, then accrual is stopped. If two of the first three patients experienced DLT, then an additional three patients could be accrued at that dose level, but dose escalation could take place only if none of the additional cohort experienced DLT. The last planned dose escalation is to 300 mg/m2. Cohorts of at least 3 patients will be entered at each dose level and monitored for at least 4 weeks after treatment before dose escalation. Intrapatient dose escalation is not permitted.

Dose level Dose of IP CPT-11(mg/m2)

1. 50
2. 100
3. 150
4. 200
5. 300

In this study, DLT is defined as follows: any grade 4 non-hematologic toxicity or as noted below; ≥ grade 3 diarrhea or stomatitis lasting ≥ 7 days despite optimal supportive care; hematologic dose-limiting toxicity is defined grade 4 neutropenia complicated by fever ≥ 38°C; grade 4 hemorrhage or thrombocytopenia; failure to recover neutrophils (≥ 1500/ mm3) or platelets (≥ 100 000/ mm3) by day 28. The maximal tolerated dose is defined as that dose level that produced dose-limiting toxicity in ≥ 50% of patients. The recommended dose is one level below that. During the study, the evaluation of toxicities will be done daily of postoperative 6 days then weekly using National Cancer Institute-Common Toxicity Criteria (NCI-CTC). Physical examination, complete blood count, and blood chemistry, and serum electrolytes will be measured. Pharmacokinetic study : Plasma, peritoneal fluid and urine samples will be assayed for irinotecan and its metabolites: SN-38, 7-ethyl-10-[4-N-(5-aminopentanoic acid)-1-piperidino] carbonyl camptothecin (APC), and SN-38 glucuronide(SN-38G).

ELIGIBILITY:
Inclusion Criteria:Patients will be eligible for the following criteria are met;

* Histologic diagnosis of gastric adenocarcinoma
* Preoperative studies of resectable disease; endoscopic finding of advanced gastric cancer, radiologic finding of T3 or T4 disease with or without suspicious peritoneal seeding
* Males or females at least 18 years of age
* Performance status 0-1 on the ECOG criteria
* The operative finding and biopsy of suspected peritoneum must show peritoneal involvement of adenocarcinoma
* No previous chemotherapy, immunotherapy or radiotherapy
* No biological major abnormalities.
* Adequate hematologic (WBC count ≥ 4,000/mm3, platelet count ≥ 150,000/mm3), hepatic (bilirubin level £ 1.5 mg/dL), and renal (creatinine concentration £ 1.5 mg/dL) function.
* Informed consent from patient or patient's relative
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards

Exclusion Criteria:

* Myocardial infarction within preceding 6 months or symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia
* Serious concomitant infection
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence)
* History of significant neurologic or psychiatric disorders
* Pregnant or lactating women
* Women of child bearing potential not using a contraceptive method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-10; Primary Completion 2006-12 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The objectives of this study are to assess the feasibility, to determine the maximum tolerated dose, and to assess the toxicities of intraperitoneally administered CPT-11 in gastric cancer patients with peritoneal seeding. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Young Suk Park, M.D.,Ph.D., Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Guichard S, Chatelut E, Lochon I, Bugat R, Mahjoubi M, Canal P. Comparison of the pharmacokinetics and efficacy of irinotecan after administration by the intravenous versus intraperitoneal route in mice. Cancer Chemother Pharmacol. 1998;42(2):165-70. doi: 10.1007/s002800050801. PMID 9654118
- [Result] Maruyama M, Nagahama T, Yuasa Y. Intraperitoneal versus intravenous CPT-11 for peritoneal seeding and liver metastasis. Anticancer Res. 1999 Sep-Oct;19(5B):4187-91. PMID 10628373
- [Result] Rosen HR, Jatzko G, Repse S, Potrc S, Neudorfer H, Sandbichler P, Zacherl J, Rabl H, Holzberger P, Lisborg P, Czeijka M. Adjuvant intraperitoneal chemotherapy with carbon-adsorbed mitomycin in patients with gastric cancer: results of a randomized multicenter trial of the Austrian Working Group for Surgical Oncology. J Clin Oncol. 1998 Aug;16(8):2733-8. doi: 10.1200/JCO.1998.16.8.2733. PMID 9704725
- [Result] Rothenberg ML, Liu PY, Braly PS, Wilczynski SP, Hannigan EV, Wadler S, Stuart G, Jiang C, Markman M, Alberts DS. Combined intraperitoneal and intravenous chemotherapy for women with optimally debulked ovarian cancer: results from an intergroup phase II trial. J Clin Oncol. 2003 Apr 1;21(7):1313-9. doi: 10.1200/JCO.2003.07.031. PMID 12663720